CLINICAL TRIAL: NCT01692379
Title: RandomizEd Trial of reVascularizAtion With Solitaire FR® Device Versus Best mediCal Therapy in the Treatment of Acute Stroke Due to anTerior Circulation Large Vessel Occlusion Presenting Within 8 Hours of Symptom Onset
Brief Title: Endovascular Revascularization With Solitaire Device Versus Best Medical Therapy in Anterior Circulation Stroke Within 8 Hours
Acronym: REVASCAT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Following DSMB advice after first interim analysis (n=174)
Sponsor: Fundacio Ictus Malaltia Vascular (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REVASCAT
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Acute Stroke
Keywords: Acute ischemic stroke; endovascular treatment; clinical trial
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endovascular treatment (Experimental): Mechanical embolectomy with Solitaire FR device
  Interventions: Device: Solitaire FR device
- Medical treatment (Active Comparator): Medical treatment (standard of care in acute ischemic stroke)including intravenous thrombolysis
  Interventions: Other: Medical treatment

INTERVENTIONS:
Device: Solitaire FR device — Mechanical embolectomy in anterior large vessel occlusion
  Arms: Endovascular treatment
Other: Medical treatment — Standard of care in acute ischemic stroke including intravenous rTPA
  Arms: Medical treatment

SUMMARY:
To evaluate the hypothesis that mechanical embolectomy with the Solitaire FR device is superior to medical management alone in achieving favorable outcome in the distribution of the modified Rankin Scale scores at 90 days in subjects presenting with acute large vessel ischemic stroke < 8 hours from symptom onset.

DETAILED DESCRIPTION:
Prospective, multi-center, randomized, controlled, open, blinded-endpoint trial with a sequential design. The randomization employs a 1:1 ratio of mechanical embolectomy with the CE MARK approved stentriever Solitaire FR® versus medical management alone. Randomization will be done under a minimization process using age, baseline NIHSS, therapeutic window and vessel occlusion site. For the primary endpoint, subjects will be followed for 90 days post-randomization.

Interim analysis will be performed as preplanned and interpreted by the Data Safety Monitoring Board (DSMB) after the first 174, 346 and 518 patients representing 25%, 50% and 75% of the planned sample size have completed their 90-day follow-up. The DSMB will advise the executive committee (EC) on recommendations to stop the trial early either for reasons of safety, efficacy, futility or to adjust the sample size. The latter may be necessary as given the paucity of data regarding natural history of the non-treated patients assumptions regarding rates of favorable outcomes in this group of patients may be incorrect. Of note, sample size adjustment based on different than expected outcomes rates is permitted, but it is not permitted to adjust the sample size based on change in the pre-specified treatment effect which is set at 10%.

Subject population: Subjects presenting with acute ischemic stroke within 8 hours from symptom onset and whose strokes are attributable to an occlusion of the internal carotid or proximal MCA (M1) arteries. Subjects are either ineligible for IV alteplase or have received IV alteplase therapy without recanalization.

ELIGIBILITY:
Inclusion Criteria:

* 1. Acute ischemic stroke where patient is ineligible for IV thrombolytic treatment or the treatment is contraindicated (e.g., subject presents beyond recommended time from symptom onset), or where patient has received IV thrombolytic therapy without recanalization after a minimum of 30 min from start of iv tPA infusion
* 2. No significant pre-stroke functional disability (mRS ≤ 1)
* 3. Baseline NIHSS score obtained prior to randomization must be equal or higher than 6 points
* 4. Age ≥18 and ≤ 85.
* 5. Occlusion (TICI 0-1) of the intracranial ICA (distal ICA or T occlusions), MCA-M1 segment or tandem proximal ICA/MCA-M1 suitable for endovascular treatment, as evidenced by CTA, MRA or angiogram, with or without concomitant cervical carotid occlusion or stenosis
* 6. Patient treatable within eight hours of symptom onset. Symptoms onset is defined as point in time the patient was last seen well (at baseline). Treatment start is defined as groin puncture.
* 7. Informed consent obtained from patient or acceptable patient surrogate

Exclusion Criteria:

* Clinical criteria
* 1. Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 3.0
* 2. Baseline platelet count < 30.000/µL
* 3. Baseline blood glucose of < 50mg/dL or >400mg/dl
* 4. Severe, sustained hypertension (SBP > 185 mm Hg or DBP > 110 mm Hg)
* 5. Patients in coma (NIHSS item of consciousness >1) (Intubated patients for transfer could be randomized only in case an NIHSS is obtained by a neurologist prior transportation).
* 6. Seizures at stroke onset which would preclude obtaining a baseline NIHSS
* 7. Serious, advanced, or terminal illness with anticipated life expectancy of less than one year.
* 8. History of life threatening allergy (more than rash) to contrast medium
* 9. Subjects who has received iv t-PA treatment beyond 4,5 hours from the beginning of the symptoms
* 10. Renal insufficiency with creatinine ≥ 3 mg/dl
* 11. Woman of childbearing potential who is known to be pregnant or lactating or who has a positive pregnancy test on admission.
* 12. Subject participating in a study involving an investigational drug or device that would impact this study.
* 13. Cerebral vasculitis
* 14. Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations, mRS score at baseline must be ≤ 1. This excludes patients who are severely demented, require constant assistance in a nursing home type setting or who live at home but are not fully independent in activities of daily living (toileting, dressing, eating, cooking and preparing meals, etc.)
* 15. Unlikely to be available for 90-day follow-up (e.g. no fixed home address, visitor from overseas).

Neuroimaging criteria:

* 16. Hypodensity on CT or restricted diffusion amounting to an ASPECTS score of <7 on NCCT or <6 on DWI MRI. Patients 81 to 85 years old with ASPECTS score on non-contrast CT or DWI MRI <9 must be excluded. ASPECTS must be evaluated by CBV maps of CT Perfusion, CTA source imaging (CTA-SI) or DWI-MR in patients whose vascular occlusion study (CTA/MRA) confirming qualifying occlusion, is performed beyond 4.5 hours of last seen well.
* 17. CT or MR evidence of hemorrhage (the presence of microbleeds is allowed).
* 18. Significant mass effect with midline shift.
* 19. Evidence of ipsilateral carotid occlusion, high grade stenosis or arterial dissection in the extracranial or petrous segment of the internal carotid artery that cannot be treated or will prevent access to the intracranial clot or excessive tortuosity of cervical vessels precluding device delivery/deployment
* 20. Subjects with occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation)
* 21. Evidence of intracranial tumor (except small meningioma).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2012-11; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Between-group comparison of the distribution of the modified Rankin Scale scores (shift analysis) | 90 days after enrollment
  evaluated by two separate assessors who are blinded to treatment

SECONDARY OUTCOMES:
Mortality at 90 days | 90 days after enrollment
Symptomatic Intracerebral Hemorrhage | 24h (-2/+12 hours) after enrollment
  Deterioration in NIHSS score of ≥4 points within 24 hours from treatment and evidence of intraparenchymal hemorrhage type 2 in the 22 to 36 hours follow-up imaging scans evaluated by independent CT/MR Core Lab and Clinical Events Committee
Infarct Volume | 24h (-2/+12h) post treatment
  Infarct volume evaluated in a second neuroimaging after treatment evaluated by independent CT/MR Core Lab
Vessel recanalization | 24h post treatment
  Vessel recanalization evaluated by CT angiography or MRA at 24 hours in both treatment groups evaluated by independent CT/MR Core Lab
Intraprocedural related complications in endovascular arm | During endovascular treatment
  Procedural related complications in the endovascular treatment arm: arterial perforation, arterial dissection, and embolization in a previously uninvolved vascular territory evaluated by the Angiography Core Lab and the Clinical Events Committee

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Dávalos, MD, Study Chair — Hospital Universitario Germans Trias i Pujol, Barcelona, Spain; Tudor Jovin, MD, Study Chair — UPMC Stroke Institute, Pittsburgh, PA, USA; Angel Chamorro, MD, Study Director — Hospital Clinic Barcelona, Barcelona, Spain; Joaquin Serena, MD, Study Director — Hospital Josep Trueta, Girona, Spain; Alex Rovira, MD, Study Director — Hospital Vall D'Hebron, Barcelona, Spain; Maria A De Miquel, MD, Study Director — Hospital de Bellvitge, Barcelona, Spain; Luis Sanromán, MD, Study Director — Hospital Clinic, Barcelona, Spain; Erik Cobo, MD, Study Director — UPC, Barcelona, Spain; Carlos Molina, MD, Study Director — Hospital Vall D'Hebron, Barcelona, Spain
Locations (4):
- Spain (4):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Vall D'Hebron, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona
  - Hospital Universitari Bellvitge, L'Hospitalet de Llobregat, Barcelona

REFERENCES:
- [Background] Molina CA, Chamorro A, Rovira A, de Miquel A, Serena J, Roman LS, Jovin TG, Davalos A, Cobo E. REVASCAT: a randomized trial of revascularization with SOLITAIRE FR device vs. best medical therapy in the treatment of acute stroke due to anterior circulation large vessel occlusion presenting within eight-hours of symptom onset. Int J Stroke. 2015 Jun;10(4):619-26. doi: 10.1111/ijs.12157. Epub 2013 Nov 10. PMID 24206399
- [Derived] Kaneko N, Komuro Y, Yokota H, Tateshima S. Stent retrievers with segmented design improve the efficacy of thrombectomy in tortuous vessels. J Neurointerv Surg. 2019 Feb;11(2):119-122. doi: 10.1136/neurintsurg-2018-014061. Epub 2018 Jul 24. PMID 30045949
- [Derived] Al-Ajlan FS, Al Sultan AS, Minhas P, Assis Z, de Miquel MA, Millan M, San Roman L, Tomassello A, Demchuk AM, Jovin TG, Cuadras P, Davalos A, Goyal M, Menon BK; REVASCAT Investigators. Posttreatment Infarct Volumes when Compared with 24-Hour and 90-Day Clinical Outcomes: Insights from the REVASCAT Randomized Controlled Trial. AJNR Am J Neuroradiol. 2018 Jan;39(1):107-110. doi: 10.3174/ajnr.A5463. Epub 2017 Nov 23. PMID 29170266
- [Derived] Davalos A, Cobo E, Molina CA, Chamorro A, de Miquel MA, Roman LS, Serena J, Lopez-Cancio E, Ribo M, Millan M, Urra X, Cardona P, Tomasello A, Castano C, Blasco J, Aja L, Rubiera M, Gomis M, Renu A, Lara B, Marti-Fabregas J, Jankowitz B, Cerda N, Jovin TG; REVASCAT Trial Investigators. Safety and efficacy of thrombectomy in acute ischaemic stroke (REVASCAT): 1-year follow-up of a randomised open-label trial. Lancet Neurol. 2017 May;16(5):369-376. doi: 10.1016/S1474-4422(17)30047-9. Epub 2017 Mar 16. PMID 28318984
- [Derived] Millan M, Remollo S, Quesada H, Renu A, Tomasello A, Minhas P, Perez de la Ossa N, Rubiera M, Llull L, Cardona P, Al-Ajlan F, Hernandez M, Assis Z, Demchuk AM, Jovin T, Davalos A; REVASCAT Trial Investigators. Vessel Patency at 24 Hours and Its Relationship With Clinical Outcomes and Infarct Volume in REVASCAT Trial (Randomized Trial of Revascularization With Solitaire FR Device Versus Best Medical Therapy in the Treatment of Acute Stroke Due to Anterior Circulation Large Vessel Occlusion Presenting Within Eight Hours of Symptom Onset). Stroke. 2017 Apr;48(4):983-989. doi: 10.1161/STROKEAHA.116.015455. Epub 2017 Mar 14. PMID 28292867
- [Derived] Lopez-Cancio E, Jovin TG, Cobo E, Cerda N, Jimenez M, Gomis M, Hernandez-Perez M, Caceres C, Cardona P, Lara B, Renu A, Llull L, Boned S, Muchada M, Davalos A. Endovascular treatment improves cognition after stroke: A secondary analysis of REVASCAT trial. Neurology. 2017 Jan 17;88(3):245-251. doi: 10.1212/WNL.0000000000003517. Epub 2016 Dec 9. PMID 27940648
- [Derived] Ribo M, Molina CA, Cobo E, Cerda N, Tomasello A, Quesada H, De Miquel MA, Millan M, Castano C, Urra X, Sanroman L, Davalos A, Jovin T; REVASCAT Trial Investigators. Association Between Time to Reperfusion and Outcome Is Primarily Driven by the Time From Imaging to Reperfusion. Stroke. 2016 Apr;47(4):999-1004. doi: 10.1161/STROKEAHA.115.011721. Epub 2016 Mar 8. PMID 26956258
- [Derived] Lopez-Cancio E, Salvat M, Cerda N, Jimenez M, Codas J, Llull L, Boned S, Cano LM, Lara B, Molina C, Cobo E, Davalos A, Jovin TG, Serena J; REVASCAT investigators. Phone and Video-Based Modalities of Central Blinded Adjudication of Modified Rankin Scores in an Endovascular Stroke Trial. Stroke. 2015 Dec;46(12):3405-10. doi: 10.1161/STROKEAHA.115.010909. Epub 2015 Nov 5. PMID 26542697
- [Derived] Urra X, Abilleira S, Dorado L, Ribo M, Cardona P, Millan M, Chamorro A, Molina C, Cobo E, Davalos A, Jovin TG, Gallofre M; Catalan Stroke Code and Reperfusion Consortium. Mechanical Thrombectomy in and Outside the REVASCAT Trial: Insights From a Concurrent Population-Based Stroke Registry. Stroke. 2015 Dec;46(12):3437-42. doi: 10.1161/STROKEAHA.115.011050. Epub 2015 Oct 27. PMID 26508752
- [Derived] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Derived] Abilleira S, Ribera A, Davalos A, Ribo M, Chamorro A, Cardona P, Molina CA, Martinez-Yelamos A, Urra X, Dorado L, Roquer J, Marti-Fabregas J, Aja L, Tomasello A, Castano C, Blasco J, Canovas D, Castellanos M, Krupinski J, Guimaraens L, Perendreu J, Ustrell X, Purroy F, Gomez-Choco M, Baiges JJ, Cocho D, Saura J, Gallofre M; Catalan Stroke Code and Reperfusion Consortium. Functional outcome after primary endovascular therapy or IV thrombolysis alone for stroke. An observational, comparative effectiveness study. Cerebrovasc Dis. 2014;38(5):328-36. doi: 10.1159/000368433. Epub 2014 Nov 21. PMID 25428822
- See also: Fundacio Ictus is a non-profit organization sponsoring REVASCAT study — http://fundacioictus.com/